CLINICAL TRIAL: NCT01526473
Title: A Phase I Study To Evaluate The Antitumor Activity And Safety Of DUKE-002-VRP(HUHER2-ECD+TM), An Alphaviral Vector Encoding The HER2 Extracellular Domain And Transmembrane Region, In Patient With Locally Advanced Or Metastatic Human Epidermal Growth Factor Receptor 2-Positive (HER2+) Cancers Including Breast Cancer
Brief Title: A Phase I Study To Evaluate The Antitumor Activity And Safety Of AVX901
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Kim Lyerly (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor-Investigator, H. Kim Lyerly, Professor of Surgery, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00034612
Record Dates: First submitted 2012-01-24; First posted 2012-02-06 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: HER2+ Cancer
Keywords: Alphavirus; Vaccine; Immunotherapy; HER2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AVX901 (Experimental): AVX901 at 4 x 108 IU intramuscularly, given every 2 weeks for a total of three doses.
  Interventions: Biological: AVX901

INTERVENTIONS:
Biological: AVX901 — Dosing will consist of AVX901 at 4 x 10E8 IU intramuscularly, given every 2 weeks for a total of three doses.
  Other Names: VRP-HER2 ECDTM

SUMMARY:
HER2 is a protein that is over expressed in 20-30% of breast cancers. It is also found associated with lung, gastric, ovarian, and pancreatic cancers. Although there are existing therapies that can target HER2, most patients will eventually experience progression of their disease even though their cancer continues to express HER2. Therefore, new approaches are needed for treating tumors that express HER2.

This clinical trial will use an investigational cancer vaccine called HER2 VRP or AVX901. The vaccine is based on a virus called Venezuelan equine encephalitis but it has been changed so it cannot cause active infection. Instead, the virus has been changed so it tells the immune system to attack cancer cells which make HER2.

The objectives of the study are to evaluate the safety of immunization with HER2 VRP in patients with advanced or metastatic malignancies that express HER2, and to test whether immunization will causes a strong immune system attack against the cancer.

DETAILED DESCRIPTION:
Metastatic breast cancer continues to account for more than 400,000 deaths yearly with HER2 positive breast cancers representing approximately one third of cases. Despite the efficacy of trastuzumab in HER2 overexpressing breast cancer, progression of metastatic disease is inevitable. Lapatinib, when combined with capecitabine, improves time to progression in those with trastuzumab resistant disease, but lapatinib resistance also develops in the majority of these patients. HER2 overexpression is also reported in lung, gastric, ovarian, and pancreatic cancers, all of which are also in need of improved treatment options. Because HER2 continues to be expressed in patients with refractory disease, using an immune-targeting approach against HER2 remains a promising strategy. A number of clinical trials have confirmed the ability of vaccines to activate T cell and antibody responses against HER2. We propose using a propagation-defective, single-cycle, RNA replicon vector system that expresses HER2 as an antigen-specific cancer vaccine in a Phase I clinical trial in patients with advanced or metastatic malignancies expressing HER2. The vaccine was prepared from an attenuated strain of an alphavirus in which 3 of the 7 viral genes were removed and replaced with a HER2 gene to create a self-amplifying RNA (replicon) that expresses large amounts of HER2. The HER2 gene used includes the extracellular domain (ECD) and transmembrane (TM) regions of HER2 but not the ICD region. The HER2 ECDTM replicon is packaged into virus-like replicon particles (VRP) by providing the alphavirus structural proteins from separate RNA molecules. When VRP are used for immunization, the VRP infect individual cells and the replicon expresses HER2 which then induces an immune response.

The primary objective of the study is to evaluate the safety of immunization with HER2 ECDTM VRP in patients with advanced or metastatic HER2-expressing malignancies. The study will also monitor immune responses to HER2. Preliminary data on tumor response rate will also be collected.

ELIGIBILITY:
Inclusion criteria

* One of the following subgroups of patients with HER2 overexpression as follows:

  (i) Histologically-confirmed breast cancer that is metastatic or locally recurrent (7th Edition of the AJCC TNM System) and measurable and/or evaluable or non-measurable by RECIST 1.1 criteria with HER2/neu overexpression by immunohistochemistry (2+,3+) or FISH+ and progressive disease despite having received at least 1 prior FDA approved HER2 targeted (e.g. trastuzumab, trastuzumab plus pertuzumab, T-DM1, or lapatinib) (determined by their physician).*

  *Prior therapy has at least one of the following stipulations:
* Patients may have received neoadjuvant or adjuvant treatment with prior trastuzumab or lapatinib treatment
* Patients have received a a trastuzumab, trastuzumab + pertuzumab, or T-DM1-based therapy for locally advanced or metastatic disease for a minimum of 9 weeks duration. Patients may have received more than 1 trastuzumab-based combination therapy.
* Patients have received a lapatinib-based therapy for locally advanced or metastatic disease for a minimum of 9 weeks duration. Patients may have received more than 1 lapatinib-based combination therapy.

(ii) Histologically-confirmed gastric, esophageal, or gastroesophageal adenocarcinoma that is metastatic or locally recurrent (7th Edition of the AJCC TNM System) and measurable or non-measurable by RECIST 1.1 criteria with HER2/neu overexpression by immunohistochemistry (2+,3+) or FISH+ and progressive disease despite having received at least 1 prior HER2 targeted therapy for a minimum of 9 weeks duration) (determined by their physician). or with previously documented HER2 over-expressing disease not being currently treated on a HER2 targeted therapy.

(iii) Other histologically confirmed metastatic (stage IV) or locally recurrent (stage III) (7th Edition of the AJCC TNM System) malignancy with HER2/neu overexpression by immunohistochemistry (2+,3+) or FISH+. Because there are no other malignancies with FDA approved HER2 targeting therapies, no prior HER2 directed therapy will be required for this subgroup. However, patients will have been required to have at least 1 line of therapy with a known survival benefit for their malignancy.

* Adults at least 18 years of age at the time of signing the Informed Consent Form;
* Written informed consent obtained from the patient prior to performing any study-related procedures, including screening visits. however, CT scans, bone scans, MUGA, Echocardiogram, EKG,and labs performed as standard of care prior to signing consent can be used to fulfill eligibility requirements if they were performed within 8 weeks of the first dose of AVX901 (for the MUGA or echocardiogram) and within 4 weeksof the first dose of study drug for the remainder of the studies
* Resolution of all toxic side effects of prior chemotherapy, radiotherapy or surgical procedures to NCI CTCAE (version 4.03) Grade ≤ 1 (with the exception of grade 2 alopecia, grade 2 neuropathy and grade 2 fatigue);
* Karnofsky performance status greater than or equal to 80% or ECOG status of 0 or 1 ;
* Adequate hematologic function: (WBC = 2500 mm3, hemoglobin > 10 mg/dl, platelets > 100,000/mm3);
* Adequate renal and hepatic function (Cr < 2.0 mg/dl; bilirubin < 2 X ULN; AST < 2.5 x ULN, ALT < 2.5 X ULN);
* Normal cardiac function defined as either a MUGA or ECHO with LVEF in normal institutional range (MUGA 50%; ECHO 55%);
* Female patients must be of non child-bearing potential or use effective contraception, e.g., use of oral contraceptives with an additional barrier method (since the study drug may impair the effectiveness of oral contraceptives), double barrier methods (diaphragm with spermicidal gel or condoms with contraceptive foam), Depo-Provera, partner vasectomy, total abstinence, and willing to continue the effective contraception method for 30 days after the last dose of AVX901;
* Ability to return to Duke University Medical Center for adequate follow-up as required by this protocol;
* Current therapy with endocrine agents (tamoxifen, raloxifene, torimifene and all aromatase inhibitors) and/or bisphosphonates and/or RANK-ligand inhibitors is permitted.

Exclusion criteria

* Except for patients on the concurrent HER2 targeted therapy (cohort 2) cohort, patients may not receive cytotoxic chemotherapy, monoclonal antibodies (other than RANK-ligand inhibitors being used for bone protection), HER2 targeted therapy such as lapatinib, or radiation therapy in the 3 weeks before the first injection, during the injection period or for at least 2 weeks after the last injection. Patients may have received prior radiation including for brain metastases.
* History of auto-immune disease such as, but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis. Prior history of autoimmune thyroiditis or vitiligo is permitted.
* Serious chronic or acute illness considered by the P.I. to constitute an unwarranted high risk for investigational drug treatment.
* Medical or psychological impediment to probable compliance with the protocol.
* Concurrent or prior second malignancy (within the past 5 years) other than non-melanoma skin cancer, controlled superficial bladder cancer or controlled cervical cancer.
* Presence of active infection or systemic use of antimicrobials within 72 hours prior to the first injection
* Patients on steroid therapy (or other immunosuppressives such as azathioprine or cyclosporine A) are excluded on the basis of potential immune suppression. Patients must have had 6 weeks of discontinuation of any steroid therapy prior to enrollment (except steroids used as anti-emetics for systemic chemotherapy which are permitted).
* Presence of an active acute or chronic infection including HIV (as determined by ELISA and confirmed by Western Blot) or viral hepatitis (as determined by HBsAg and Hepatitis C serology). Patients with HIV are excluded based on immuno-suppression, which may render them unable to respond to the vaccine; patients with chronic hepatitis are excluded because of concern that hepatitis could be exacerbated by the injections. .
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Safety | 3 months
  The primary objective of the study is to evaluate the safety of immunization with HER2 ECDTM VRP in patients with advanced or metastatic HER2-expressing malignancies

SECONDARY OUTCOMES:
Immune response | 3 months
  The secondary objective of the study HER2 specific response by ELISPOT and ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morse, MD, Principal Investigator — Duke University; H. Kim Lyerly, MD, Study Director — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States